CLINICAL TRIAL: NCT01004003
Title: A Multicenter, Open Label, Phase I /Randomised Phase II Study to Evaluate Safety, Pharmacokinetics and Efficacy of BIBF 1120 in Comparison With Oral Sorafenib for Advanced Hepatocellular Carcinoma Patients.
Brief Title: Phase I/II Comparison of Efficacy and Safety of BIBF 1120 and Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.37; 2009-011925-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-10-12; First posted 2009-10-29 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; nintedanib

ARMS (2):
- BIBF 1120 (Experimental): Phase I dose escalation and phase II using dose determined in phase I ( 200 mg BID)
  Interventions: Drug: BIBF 1120
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib
  Arms: Sorafenib
Drug: BIBF 1120 — Dose escalated in phase I until MTD or adjusted by investigator, dose in phase II part based on phase I data
  Arms: BIBF 1120

SUMMARY:
The study aim is to determine maximally tolerated dose (MTD) of BIBF 1120 in HCC (hepatocellular cancer) and compare efficacy of BIBF 1120 to Sorafenib in HCC patients

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of hepatocellular carcinoma (HCC) not amenable to curative surgery or loco-regional therapy (RFA, percutaneous ethanol injection (PEI), TACE)
* Age 18 years or older
* Eastern Cooperative Oncology Group performance score of 2 or less
* Child-Pugh score A (score 5-6)
* At least one measurable lesion according to RECIST 1.0 (this criterion is limited to phase II only)
* In case a measurable lesion was previously treated by loco-regional therapy (RFA, PEI, TACE or RT) , this lesion must have to be documented as progression according to RECIST 1.0 by CT or MRI (this criterion is limited to phase II only).
* Time interval from last local therapy (e.g. radiofrequency ablation, percutaneous ethanol injection, radiotherapy, transarterial chemoembolization) more than 4 weeks prior to start of study treatment
* Written informed consent consistent with International Conference on Harmonisation/ Good Clinical Practice (ICH-GCP) and local legislation

Exclusion criteria:

* Prior systemic therapy for HCC
* Fibrolamellar hepatocellular carcinoma (HCC)
* Bilirubin greater than 1.5 times ULN
* AST or ALT greater than 2 times ULN
* Uncontrolled or refractory ascites to adequate medical therapy
* Hepatic encephalopathy more than grade 1 according to Child-Pugh criteria
* Prothrombin time international normalized ratio greater than 2.3, or prothrombin time more than 6 seconds prolonged than control
* Absolute neutrophil count less than 1000 /µL
* Platelet count less than 60000 /µL
* Hemoglobin less than 9 g/dL
* Serum creatinine greater than 1.5 times Upper Limit of Normal (ULN)
* Proteinuria of Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or greater
* Variceal bleeding within last 6 months prior to start of study treatment
* History of major thrombotic (except portal vein thrombosis) or clinically relevant major bleeding event in the past 6 months
* Known inherited predisposition to bleeding or thrombosis
* Significant cardiovascular diseases (i.e. hypertension not controlled by medical therapy, blood pressure > 150/90 mmHg), unstable angina, history of myocardial infarction within the past 6 months, congestive heart failure > class II according to New York Heart Association (NYHA), serious cardiac arrhythmia, pericardial effusion)
* Therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except for chronic low-dose therapy with acetylsalicylic acid =< 325mg per day)
* Major surgery within 4 weeks prior to start of study treatment
* Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
* Known serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least twelve months after end of active therapy
* Current alcohol abuse or drug abuse that would limit pt ability to comply with protocol
* Symptomatic central nervous system (CNS) metastasis
* Life expectancy less than 12 weeks
* Patient unable to take oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-10-22 (Actual); Primary Completion 2014-07-14 (Actual); Study Completion 2016-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (28):
- Austria (2):
  - 1199.37.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1199.37.43002 Boehringer Ingelheim Investigational Site, Vienna
- France (2):
  - 1199.37.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1199.37.33002 Boehringer Ingelheim Investigational Site, Paris
- Germany (9):
  - 1199.37.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 1199.37.49009 Boehringer Ingelheim Investigational Site, Erlangen
  - 1199.37.49002 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1199.37.49001 Boehringer Ingelheim Investigational Site, Hanover
  - 1199.37.49010 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1199.37.49005 Boehringer Ingelheim Investigational Site, Jena
  - 1199.37.49004 Boehringer Ingelheim Investigational Site, Magdeburg
  - 1199.37.49003 Boehringer Ingelheim Investigational Site, München
  - 1199.37.49006 Boehringer Ingelheim Investigational Site, Tübingen
- 1199.37.36001 Boehringer Ingelheim Investigational Site, Debrecen, Hungary
- Netherlands (2):
  - 1199.37.31002 Boehringer Ingelheim Investigational Site, Leiden
  - 1199.37.31001 Boehringer Ingelheim Investigational Site, Utrecht
- Poland (3):
  - 1199.37.48002 Boehringer Ingelheim Investigational Site, Olsztyn
  - 1199.37.48001 Boehringer Ingelheim Investigational Site, Warsaw
  - 1199.37.48003 Boehringer Ingelheim Investigational Site, Warsaw
- Romania (2):
  - 1199.37.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1199.37.40003 Boehringer Ingelheim Investigational Site, Cluj-Napoca
- United Kingdom (7):
  - 1199.37.44001 Boehringer Ingelheim Investigational Site, Edgbaston, Birmingham
  - 1199.37.44005 Boehringer Ingelheim Investigational Site, Glasgow
  - 1199.37.44008 Boehringer Ingelheim Investigational Site, Liverpool
  - 1199.37.44002 Boehringer Ingelheim Investigational Site, London
  - 1199.37.44003 Boehringer Ingelheim Investigational Site, London
  - 1199.37.44006 Boehringer Ingelheim Investigational Site, Manchester
  - 1199.37.44004 Boehringer Ingelheim Investigational Site, Nottingham

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Group 1, 100mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid). Phase I: A standard 3+3 dose escalation part to determine the maximal tolerated dose (MTD). Group 1 patients had a baseline Child-Pugh score of 5 or 6, and aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤2 times the upper limit of normal (ULN).
- Phase I Group 1, 150mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 150 mg soft gelatine capsules twice daily (bid). Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 1 patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN).
- Phase I Group 1, 200mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules (two capsules of 100mg) twice daily (bid). Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 1 patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN).
- Phase I Group 2, 50mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 50 mg soft gelatine capsules twice daily (bid). Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
- Phase I Group 2, 100mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid). Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
- Phase I Group 2, 150mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 150 mg soft gelatine capsules twice daily (bid). Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
- Phase I Group 2, 200mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules (two capsules of 100mg) twice daily (bid). Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
- Phase II, 200 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules (two capsules of 100mg) twice daily (bid). Phase II: Patients were randomly assigned to open-label treatment with nintedanib or sorafenib. Patients were stratified for macrovascular invasion (MVI) and/or extra-hepatic spread (EHS). Patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN).
- Phase II, 400 mg Sorafenib Bid: Oral administration of Sorafenib 400 mg film coated tablets twice daily (bid). Phase II: Patients were randomly assigned to open-label treatment with nintedanib or sorafenib. Patients were stratified for macrovascular invasion (MVI) and/or extra-hepatic spread (EHS). Patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN).
Period: Overall Study
Arm/Group | Phase 1 Group 1, 100mg Nintedanib Bid | Phase I Group 1, 150mg Nintedanib Bid | Phase I Group 1, 200mg Nintedanib Bid | Phase I Group 2, 50mg Nintedanib Bid | Phase I Group 2, 100mg Nintedanib Bid | Phase I Group 2, 150mg Nintedanib Bid | Phase I Group 2, 200mg Nintedanib Bid | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Started | 6 | 3 | 4 | 3 | 4 | 4 | 8 | 62 | 31
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (On-treatment at analysis cut-off date (15 July 2014).) | 1 (On-treatment at analysis cut-off date (15 July 2014).)
Not Completed | 6 | 3 | 4 | 3 | 4 | 4 | 8 | 60 | 30
Not completed — Progressive disease | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 39 | 22
Not completed — Adverse Event | 4 | 2 | 3 | 3 | 2 | 2 | 7 | 21 | 6
Not completed — Refused to continue taking trial med. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients who received at least one single dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Group 1, 100mg Nintedanib Bid | Phase I Group 1, 150mg Nintedanib Bid | Phase I Group 1, 200mg Nintedanib Bid | Phase I Group 2, 50mg Nintedanib Bid | Phase I Group 2, 100mg Nintedanib Bid | Phase I Group 2, 150mg Nintedanib Bid | Phase I Group 2, 200mg Nintedanib Bid | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid | Total
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 4 | 4 | 8 | 62 | 31 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (6.8) | 65.0 (7.8) | 66.5 (4.0) | 72.3 (11.7) | 56.3 (6.4) | 59.3 (13.9) | 57.0 (11.0) | 65.4 (10.0) | 63.1 (11.8) | 64.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 14 | 5 | 24
  Male | 5 | 2 | 4 | 3 | 4 | 3 | 6 | 48 | 26 | 101

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose in Phase I
Description: The MTD was defined as the highest dose studied for which the incidence of dose limiting toxicities (DLTs) was 0/3 or less than 2/6 patients during the first treatment course.
Time Frame: 4 weeks
Population: Treated set which included all patients who received at least one single dose of trial medication, including phase I patients from the dose escalation part that were not replaced for MTD determination.
Measure: Number; unit: mg bid
Groups:
- Group 1: Patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN)
- Group 2: Patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 13
mg bid | 200 | 200

2. Primary Outcome: Time to Progression (TTP) in Phase II
Description: TTP according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.0 criteria based on central independent review. TTP RECIST 1.0 was defined as the time from randomisation to disease progression according to RECIST 1.0.
Time Frame: From randomization until data cut-off (15 July 2014); Up to 1031 days
Population: Treated set, only phase II participants.
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Phase II, 400 mg Sorafenib Bid: Oral administration of Sorafenib 400 mg film coated tablets twice daily (bid). Phase II: Patients were randomly assigned to open-label treatment with nintedanib or sorafenib. Patients were stratified for macro-vascular invasion (MVI) and/or extra-hepatic spread (EHS). Patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN).
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 62 | 31
months | 5.45 [2.69 to 9.20] | 4.63 [2.79 to 20.40]
Statistical Analysis 1: Comparison: Phase II, 200 mg Nintedanib Bid vs Phase II, 400 mg Sorafenib Bid; Test type: Superiority or Other; Hazard Ratio (HR) = 1.437, 95% CI 2-sided [0.805 to 2.565] — Hazard ratio (HR) from Cox proportional hazards model stratified by macroscopic vacular invasion, extrahepatic spread, or both present vs both absent. HR below 1 favors Nintedanib

3. Secondary Outcome: Incidence of Dose Limiting Toxicity in Phase I
Description: Number of patients with dose limiting toxicity are presented
Time Frame: 4 weeks
Population: Treated set (Phase I patients from the dose escalation part that were not replaced for MTD determination).
Measure: Number; unit: participants
Groups:
- Phase I Group I, 100 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the maximal tolerated dose (MTD).
  Group 1 patients had a baseline Child-Pugh score of 5 or 6, and AST (aspartate aminotransferase ) and ALT (alanine transaminase) ≤2 times the upper limit of normal (ULN).
- Phase I Group 1, 150 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 150 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 1 patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN).
- Phase I Group 1, 200 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules (two capsules of 100mg) twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 1 patients had a baseline Child-Pugh score of 5 or 6, and AST and ALT ≤2 times the upper limit of normal (ULN).
- Phase I Group 2, 50 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 50 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
- Phase I Group 2, 100 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
- Phase I Group 2, 150 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 150 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
- Phase I Group 2, 200 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules (two capsules of 100mg)twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD. Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN.
Arm/Group | Phase I Group I, 100 mg Nintedanib Bid | Phase I Group 1, 150 mg Nintedanib Bid | Phase I Group 1, 200 mg Nintedanib Bid | Phase I Group 2, 50 mg Nintedanib Bid | Phase I Group 2, 100 mg Nintedanib Bid | Phase I Group 2, 150 mg Nintedanib Bid | Phase I Group 2, 200 mg Nintedanib Bid
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Objective Tumour Response by RECIST
Description: Objective RECIST 1.0 tumour response was defined as Complete Response (CR) or Partial Response (PR) and was derived from the patient's best objective RECIST 1.0 response based on central independent review.
  95% Confidence Interval presented below are computed by Clopper and Pearson method.
Time Frame: From randomization until data cut-off (15 July 2014); Up to 1031 days
Population: Treated set, phase II participants only
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 62 | 31
percentage of participants | 1.6 [0.0 to 8.7] | 6.5 [0.8 to 21.4]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS by RECIST 1.0 was defined as the duration from date of randomisation to date of progression or death, whichever occurred earlier, based on central independent review.
Time Frame: From randomization until data cut-off (15 July 2014); Up to 1031 days
Population: Treated set, only phase II participants
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 62 | 31
months | 5.32 [2.69 to 9.20] | 3.94 [2.33 to 7.36]
Statistical Analysis 1: Comparison: Phase II, 200 mg Nintedanib Bid vs Phase II, 400 mg Sorafenib Bid; Test type: Superiority or Other; Hazard Ratio (HR) = 1.351, 95% CI 2-sided [0.779 to 2.343] — Hazard ratio from Cox proportional hazards model stratified by macroscopic vacular invasion, extrahepatic spread, or both present vs both absent. HR below 1 favors Nintedanib

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the duration from date of randomisation to the date of death.
Time Frame: From randomization until data cut-off (15 July 2014); Up to 1031 days
Population: Treated set, only phase II participants
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 62 | 31
months | 11.86 [6.60 to 25.46] | 11.40 [6.51 to 17.25]
Statistical Analysis 1: Comparison: Phase II, 200 mg Nintedanib Bid vs Phase II, 400 mg Sorafenib Bid; Test type: Superiority or Other; Hazard Ratio (HR) = 0.877, 95% CI 2-sided [0.522 to 1.473] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: From first administration of the trial drug and until 28 days after the last administration of nintedanib or sorafenib, up to 1289 days
Arm/Group | Phase 1 Group 1, 100mg Nintedanib Bid | Phase I Group 1, 150mg Nintedanib Bid | Phase I Group 1, 200mg Nintedanib Bid | Phase I Group 2, 50mg Nintedanib Bid | Phase I Group 2, 100mg Nintedanib Bid | Phase I Group 2, 150mg Nintedanib Bid | Phase I Group 2, 200mg Nintedanib Bid | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/3 | 4/4 | 3/3 | 2/4 | 3/4 | 4/8 | 34/62 | 14/31
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 4/4 | 3/3 | 4/4 | 4/4 | 7/8 | 61/62 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Group 1, 100mg Nintedanib Bid (N=6) | Phase I Group 1, 150mg Nintedanib Bid (N=3) | Phase I Group 1, 200mg Nintedanib Bid (N=4) | Phase I Group 2, 50mg Nintedanib Bid (N=3) | Phase I Group 2, 100mg Nintedanib Bid (N=4) | Phase I Group 2, 150mg Nintedanib Bid (N=4) | Phase I Group 2, 200mg Nintedanib Bid (N=8) | Phase II, 200 mg Nintedanib Bid (N=62) | Phase II, 400 mg Sorafenib Bid (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ludwig angina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 3
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Group 1, 100mg Nintedanib Bid (N=6) | Phase I Group 1, 150mg Nintedanib Bid (N=3) | Phase I Group 1, 200mg Nintedanib Bid (N=4) | Phase I Group 2, 50mg Nintedanib Bid (N=3) | Phase I Group 2, 100mg Nintedanib Bid (N=4) | Phase I Group 2, 150mg Nintedanib Bid (N=4) | Phase I Group 2, 200mg Nintedanib Bid (N=8) | Phase II, 200 mg Nintedanib Bid (N=62) | Phase II, 400 mg Sorafenib Bid (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2 | 1 | 1 | 0 | 3 | 15 | 9
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 16 | 4
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anorectal varices (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3 | 3 | 2 | 3 | 5 | 43 | 21
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 2 | 1 | 3 | 7 | 29 | 9
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 3 | 2 | 2 | 1 | 5 | 23 | 9
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Catheter site bruise (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Device difficult to use (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 3 | 2 | 1 | 2 | 5 | 32 | 10
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 8 | 1
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 10 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 3
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 6 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 3
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 2
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 8 | 3
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 11 | 5
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 6 | 2
Blood bilirubin increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 8 | 6
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 8 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 2 | 2 | 5 | 23 | 13
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 6 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 6 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 4 | 3
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 8 | 5
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 5 | 8
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 2 | 0 | 2 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 7 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 11
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 9 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 6 | 7
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 7 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Intra-abdominal haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.